CLINICAL TRIAL: NCT06043180
Title: Observational Study of Outcome Prediction in Patients Undergoing Transcatheter Aortic Valve Implantation (TAVI) for Severe Symptomatic Aortic Stenosis (PREDICT-TAVI).
Brief Title: Outcome Prediction in Patients With Aortic Stenosis After TAVI
Acronym: PREDICT-TAVI
Status: Not yet recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 319698
Record Dates: First submitted 2023-05-23; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-05

CONDITIONS: Aortic Stenosis, Severe
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe aortic stenosis: Aortic valve area <1.0 cm2/<0.6cm2/m2 or mean gradient >40mmHg or jet velocity >4.0 m/s.
  Interventions: Procedure: Transcatheter aortic valve implantation

INTERVENTIONS:
Procedure: Transcatheter aortic valve implantation — Intervention on aortic valve for severe aortic stenosis

SUMMARY:
This study will investigate changes right ventricular function and functional recovery metrics after transcatheter aortic valve implantation

DETAILED DESCRIPTION:
Aortic stenosis (AS), is a condition in which the aortic valve becomes narrowed as people get older, causing the heart pump (the left ventricle) to struggle to push blood through it, leading to breathlessness, chest pain and blackouts. If left untreated, the prognosis is bleak (similar to lung cancer). Previously the only effective treatment for AS was a valve replacement via open heart surgery, which was too high risk for many patients to undergo, meaning they were left without treatment. Over the last decade transcatheter aortic valve implantation (TAVI) has emerged as a treatment option for most patients with severe symptomatic AS. In TAVI, a new valve is inserted through a small tube, usually in the leg artery, which avoids open heart surgery.

Clinical outcomes after TAVI have significantly improved with the accumulation of operator and institution experience as well as the wide use of newer generation devices. However, a significant minority of patients undergoing TAVI derive little or no benefit from the procedure. Nearly a third describe no improvement in quality of life, or die within the first year. To combat this problem, it is essential we develop more sophisticated means of predicting adverse outcomes related to TAVI, to improve the selection of patients and identify patients where the potential benefit of the procedure is outweighed by unfavourable outcomes.

Assessment of physical recovery and improvement of symptoms and quality of life after TAVI is an important aspect of examining the outcomes of treatment. This is often a more meaningful and relevant treatment goal in the TAVI cohort than 'hard' clinical outcomes (like death and stroke) alone. Traditionally, less emphasis has been put on the assessment of the right side of the heart (the right ventricle) in evaluating physical recovery after TAVI.

We propose prospective observational study to evaluate the significance of the right side of the heart on the clinical outcomes related to functional recovery in patients undergoing TAVI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic severe aortic stenosis (AVA <1.0 cm2/<0.6cm2/m2 or mean gradient >40mmHg or jet velocity >4.0 m/s).

Exclusion Criteria:

* Extracardiac limitations of ambulatory exercise, cardiac rehab opt out, non-transfemoral TAVI, haemodynamic instability/cardiogenic shock, LVEF <40%, poorly controlled AF, severe COPD, primary pulmonary hypertension, evidence of cardiac amyloid, more than moderate concomitant valvular heart disease other than aortic stenosis, previous sternotomy, permanent pacemaker implant, patients enrolled in another study where participation would involve deviation from either protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients planned for transcatheter aortic valve implantation.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in TAPSE/PASP coupling measure | Baseline to immediately following intervention and 3 months follow up
  RV-PA coupling is measured using ratio of TAPSE/PASP on transthoracic echocardiography.
Change in daily accelerometer measured activity (steps) | Baseline to 3 months follow up
  Recorded on a wrist-worn accelerometer continuously for 14 days.

SECONDARY OUTCOMES:
Change in New York Heart Association (NYHA) Functional Class | Baseline to 3 months follow up
  The New York Heart Association (NYHA) Classification provides a simple way of classifying the extent of heart failure. It classifies patients in one of four categories based on their limitations during physical activity: Class I - No symptoms and no limitation in ordinary physical activity Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity. Class III - Marked limitation in activity due to symptoms Class IV - Severe limitations.
Change in N-terminal Prohormone of Brain Natriuretic Peptide (NT-proBNP Levels) | Baseline to 3 months follow up
  Biomarker of myocardial strain
Change in right ventricular efficiency as measured by ventricular arterial coupling | Baseline to immediately following intervention
  VA coupling is calculated by the ratio of effective arterial elastance (Ea), a measure of afterload, to LV end systolic elastance (Ees), a relatively load independent measure of LV chamber performance. Both these measures are expressed in mmHg/ml and as continuous variables.
Change in right ventricular strain/PASP coupling measure | Baseline to immediately following intervention and 3 months follow up
  RV-PA coupling can be measured using ratio of right ventricular strain/PASP on transthoracic echocardiography.
Change in right ventricular end-systolic volume/stroke volume coupling measure | Baseline to immediately following intervention and 3 months follow up
  RV-PA coupling can be measured using ratio of right ventricular ESV/SV on transthoracic echocardiography.
Change in right ventricular ejection fraction/PASP coupling measure | Baseline to immediately following intervention and 3 months follow up
  RV-PA coupling can be measured using ratio of right ventricular EF/PASP on transthoracic echocardiography.
Change in right ventricular S'/PASP coupling measure | Baseline to immediately following intervention and 3 months follow up
  RV-PA coupling can be measured using ratio of S'/PASP on transthoracic echocardiography.
Change in Six Minute Walk Test (6MWT Distance or 6MWD) | Baseline to 3 months follow up
  The Six Minute Walk Test (6MWT) is a practical simple test that requires a 100-ft hallway but no exercise equipment or advanced training for technicians. This test measures the distance that a patient can quickly walk ona flat, hard surface in a period of 6 minutes (the 6MWD). It evaluates the global and integrated responses of all the systems involved during exercise, including the pulmonary and cardiovascular systems, systemic circulation,peripheral circulation, blood, neuromuscular units, and muscle metabolism. It does not provide specific information on the function of each of the different organs and systems involved in exercise or the mechanism of exercise limitation, as is possible with maximal cardiopulmonary exercise testing. The self-paced 6MWT assesses the submaximal level of functional capacity.
Change in Quality of Life (QoL) as Measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ) | Baseline to 3 months follow up
  The Kansas City Cardiomyopathy Questionnaire is a 23-item, self administered instrument that quantifies physical function, symptoms, social function, self-efficacy and knowledge, and quality of life. with a range of possible subscale scores from 0 to 100, with 100 representing the least burden of symptoms. The KCCQ tool quantifies the following six (6) distinct domains and two (2) summary scores: KCCQ Symptom Domain, KCCQ Physical Function Domain, KCCQ Quality of Life Domain, KCCQ Social Limitation Domain, KCCQ Self-efficacy Domain, KCCQ Symptom Stability Domain, Clinical Summary Score and Overall Summary Score. Clinical Summary Score includes total symptom and physical function scores to correspond with NYHA Classification. Overall Summary Score includes the total symptom, physical function, social limitations and quality of life scores.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Redwood, Principal Investigator — King's College London
Locations (1):
- Guy's & St Thomas' NHS Foundation Trust, St Thomas' Hospital, London, United Kingdom